CLINICAL TRIAL: NCT06788587
Title: Exploring Feasibility and Acceptability of Prolonged Administration of High-Dose Stimulants in People With Methamphetamine Use Disorder: An Extension of a Randomized, Placebo-Controlled Trial
Brief Title: Feasibility of Long-term, High-dose Stimulant for Methamphetamine Use Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Ministere de la Sante et des Services Sociaux (Other); Health Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025_12643
Record Dates: First submitted 2025-01-10; First posted 2025-01-23 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-07

CONDITIONS: Methamphetamine Abuse; Methamphetamine-dependence; Addiction; Substance Abuse; Methamphetamine Use Disorder
Keywords: Substance use disorder; Amphetamines; Methamphetamine; Lisdexamfetamine; Treatment; Agonist therapy; Feasibility
MeSH Terms: conditions — Behavior, Addictive; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Single-centre, 2-arm, randomized, double-blind, dose-ascending, placebo-controlled extension trial. Participants will be enrolled into one of 2 treatment arms:
  * Arm 1: LDX-01 + TAU
  * Arm 2: Placebo + TAU
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LDX-01 + TAU (Experimental): Participants will receive TAU at the clinic as well as once daily over-encapsulated LDX-01 orally for 25 weeks.
  Interventions: Drug: LDX-01 plus TAU
- Placebo + TAU (Placebo Comparator): Participants will receive TAU at the clinic as well as once daily LDX-01-matched placebo orally for 25 weeks.
  Interventions: Drug: Placebo plus TAU

INTERVENTIONS:
Drug: LDX-01 plus TAU — Participants receive once daily LDX-01 for 25 weeks, as well as TAU at a clinical site. Medication is provided in 3 phases:
  Week 1 (Induction Phase): 100 mg (Days 1 and 2), 150 mg (Days 3 and 4), 200 mg (Days 5, 6 and 7); Weeks 2-21 (Maintenance Phase): 250 mg (or the maximum tolerated for each individual) ; Weeks 22-25 (Taper Phase): 200 mg (Week 22), 150 mg (Week 23), 100 mg (Week 24) and 50 mg (Week 25).
  Arms: LDX-01 + TAU
Drug: Placebo plus TAU — Participants receive once daily LDX-01-matched placebo for 25 weeks, as well as TAU at a clinical site. Medication is provided in 3 phases:
  Week 1 (Induction Phase): 100 mg (Days 1 and 2), 150 mg (Days 3 and 4), 200 mg (Days 5, 6 and 7); Weeks 2-21 (Maintenance Phase): 250 mg (or the maximum tolerated for each individual) ; Weeks 22-25 (Taper Phase): 200 mg (Week 22), 150 mg (Week 23), 100 mg (Week 24) and 50 mg (Week 25).
  Arms: Placebo + TAU

SUMMARY:
Methamphetamine use disorder (MUD) is becoming an increasing public health concern in Canada. While the evidence on the efficacy and safety of prescription psychostimulants for the treatment of MUD is promising, the knowledge on the maintenance therapy using stimulant agonist therapy is scarce and needs further investigation, especially in terms of long-term retention in treatment.

The goal of this clinical trial is to evaluate the feasibility of a long-term (25 weeks) administration of high-dose stimulant agonist therapy, using Lisdexamfetamine (LDX-01) on top of treatment-as-usual (TAU), in a population of people with moderate to severe MUD, as measured by study retention, treatment retention, treatment adherence and satisfaction compared against a placebo group.

Participants will be placed randomly into one of two groups:

1. TAU and high-dose LDX-01
2. TAU and placebo

DETAILED DESCRIPTION:
This trial is a single-centre, randomized double-blind (LDX-01), dose-ascending, placebo-controlled trial. This study is an extension to a parent trial, Addition of high-dose stimulant and engagement-focused contingency management, alone and in combination, to treatment as usual for the management of methamphetamine use disorder (ASCME): a pan-Canadian multi-centre, randomized, controlled trial (NCT05854667). Participants will be enrolled in one of the 2 treatment arms:

Arm 1 : TAU plus high-dose LDX-01 Arm 2 : TAU plus placebo

The trial will enroll 62-80 participants who have completed the parent trial in the Quebec site. The participants will be enrolled in the trial for 30 weeks.

Participation includes the following:

1. Participants will receive medication or placebo weekly for 25 weeks
2. Participants will attend the clinic for weekly treatment
3. Participants will attend the clinic once every week for study visits. At these visits, participants will be asked to provide a urine sample (Weeks 1-25: every two weeks, week 26 and week 30) and/or complete questionnaires

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 55 years of age at enrollment in the parent ASCME trial;
2. Diagnosed with a moderate to severe MUD as defined by the DSM-5 criteria;
3. Enrolled in the parent ASCME trial and completed the study up to and including the end of study visit at Week 20, Day 1;
4. Interested in avoiding relapse, decreasing methamphetamine use, or abstaining from methamphetamine use;
5. Presence of ongoing substance use, craving, or significant risk of relapse that according to the study physician, warrants extended treatment for MUD;
6. If female:

   * Be of non-childbearing potential, defined as (i) postmenopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age); or (ii) documented surgically sterilized (i.e., tubal ligation, hysterectomy, or bilateral oophorectomy); or
   * Be of childbearing potential, have a negative pregnancy test at screening, and agree to use an acceptable method of birth control throughout the study;
7. Willing to be randomized to one of 2 study arms and followed for the duration of the trial;
8. Able to start the study intervention within 28 days after completing the ASCME main trial (study no. CRISM-002);
9. Able to provide informed consent;
10. Willing to comply with study procedures;
11. Able to communicate in English or French

Exclusion Criteria:

1. Symptomatic or advanced cardiovascular disease (e.g., advanced arteriosclerosis), moderate hypertension; confirmed current hyperthyroidism; known hypersensitivity or idiosyncrasy to the sympathomimetic amines or glaucoma or any disabling, severe, or unstable medical condition (including electrolyte disturbances) that, in the opinion of the study physician, precludes safe participation or the ability to provide fully informed consent;
2. Any severe or unstable co-morbid substance use disorder that, in the opinion of the study physician, precludes safe participation in the study;
3. Participants with Opioid Use Disorder (OUD) who have been on Opioid Agonist Treatment (OAT) for <12 weeks, and not yet at stabilization dose, or at stabilization dose <4 weeks;
4. Current or a history of any serious psychiatric disorder (e.g., bipolar disorder, pre-existing psychosis, schizophrenia) that, in the opinion of the study physician, precludes safe participation in the study;
5. History of a SAE, hypersensitivity or known allergic reaction to LDX-01 or other amphetamine drugs, or hypersensitivity to the sympathomimetic amines;
6. Pregnant, nursing, or planning to become pregnant during the study period;
7. Planned extended absence during the study period (e.g., pending legal action, surgery, incarceration, inpatient residential program) in the opinion of the study physician that might prevent completion of the study;
8. Use of an investigational drug for stimulant use disorder during the 30 days before screening, confirmed via self-report or pharmacy records; excluding the use of study medication in the parent ASCME trial;
9. Use of prescribed amphetamine-type medication or medication for the treatment of stimulant use disorder (e.g., methylphenidate, modafinil, bupropion, or mirtazapine) in the 4 weeks before screening;
10. Current or anticipated need for treatment with any medication that may interact with LDX-01 (e.g., monoamine oxidase inhibitors [MAOIs]) used currently or within the past 14 days and that would preclude study participant at the discretion of the study physician;
11. ECG measurement (Bazett method for the correction of QT interval) that indicates a prolonged QTc interval (≥460 milliseconds for females and ≥450 milliseconds for males) at screening;
12. Any SAEs related to the study product in the parent trial phase that, in the opinion of the study physician, precludes safe participation in the extension study;
13. Any compliance issues related to the study product and/or study procedures during the parent trial phase that, in the opinion of the study physician, precludes safe participation in the extension study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Retention in treatment | Weeks 18, 19, 20, 21 and weeks 22, 23, 24, 25
  Retention in treatment will be measured as the proportion of study participants who receive any intervention during the 4 weeks before week 22 and 4 weeks before week 26
Treatment satisfaction | Weeks 22, 26
  Participant treatment satisfaction will be measured by evaluating participant satisfaction using the Client Satisfaction Questionnaire-8 (CSQ-8) questionnaire. The total score ranges from 8 (minimum) to 32 (maximum) with the higher values showing greater satisfaction.
Retention in study | Weeks 22, 26 and 30
  Retention in study will be measured as 1) the proportion of study participants who return for the study visit at week 22 with or without receiving the study interventions, 2) the proportion of study participants who return for the study visit at week 26 with or without receiving the study interventions, and 3) the proportion of study participants who return for the last study visit at week 30 with or without receiving the study interventions.
Treatment adherence | from week 1 day 1 to week 25
  Treatment adherence will be first, measured individually, as the total proportion of the number of the assigned medications (LDX-01/placebo) taken through the intervention (from baseline until the end of week 25) and then averaged across all study completers.

OTHER OUTCOMES:
Safety events | up to 30 weeks : from the date of enrollment until week 30
  Safety of long-term high-dose LDX-01 will be assessed through the collection of adverse event (AEs) and serious adverse event (SAEs). The number and proportions of each AE, SAE, adverse drug reaction (ADR), and unexpected ADR will be recorded weekly. For calculations, each participant's safety-related event will be counted once under the maximum severity or the strongest recorded causal relationship to study medication
QTc measurement | Screening, weeks 1, 2, 3, 7 and 22
  QTc will be measured using ECG; incidence of borderline prolonged (460-479 milliseconds for females and 450-469 milliseconds for males) and prolonged ( ≥ 480 milliseconds for females and ≥ 470 milliseconds for males) QTc interval will be measured using the Bazett method for the correction of QT interval.
Self-reported methamphetamine use | Baseline, week 1 day 1, weeks 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 26 and 30
  Self-reported methamphetamine use, is measured using the self-reported number of days of methamphetamine use during the 29 weeks of the study using the Timeline Follow Back (TLFB) Questionnaire since the last study visit, or in the past 28 days, whichever number of days is the least (i.e., researcher-administered, with memory cues to improve accuracy).
Methamphetamine use by urinalysis | week 1 day 1, weeks 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, 26 and 30
  Methamphetamine use by urinalysis will be measured by the number of reactive urine samples tested for methamphetamine using the rapid chromatographic immunoassays for urine drug screen (UDS). All urine specimens will be collected and analyzed using a Rapid Response Multi- Drug One Step Screen Test Panel, following the manufacturer's recommended procedures to test for the presence of the following drugs or their respective metabolites: methamphetamine, morphine, fentanyl, benzodiazepines, cocaine, THC, methadone, buprenorphine, methylphenidate, MDMA, LSD, ketamine, oxycodone, heroin, Hydromorphone and amphetamine (week 30 only). A validity check will be performed using an adulterant strip included in the test.
Amphetamine craving | week 1 day 1, weeks 12, 22, 26 and 30
  Amphetamine craving will be measured using the Brief Substance Craving Scale (BSCS). The BSCS is a 16-item, self-report instrument which assesses cravings for substances over 24-hour period. It has good psychometric properties. Intensity, frequency, and length of cravings are recorded on a five-point Likert scale. the total score is 0 (minimum) to 12 (maximum) with higher values indicating a larger craving.
Addiction severity | week 1 day 1, weeks 12, 22, 26 and 30
  Addiction severity is measured with the Addiction Severity Index (ASI), a Self-Report questionnaire that captures substance abuse participants' functioning. It has good psychometric properties, with good consistency and test-retest reliabilities. The ASI Self-Report assesses problem use in the past 30 days in seven areas commonly affected by substance use, including medical, employment/support, alcohol, drug, legal, family/social, and psychiatric drug sections.
Quality of life | week 1 day 1, weeks 12, 22, 26 and 30
  Quality of life will be measured using the World Health Organization Quality of Life - BREF (WHOQOL-BREF), a person-centred generic patient-reported quality of life measure, validated to document and follow changes in quality of life in different physical and psychiatric disorders. It specifically looks at 4 domains related to quality of life: physical health, psychological health, social relationships, and environment. Domain scores for the WHOQOL-BREF are calculated by taking the mean of all items included in each domain and multiplying by a factor of four. These scores are then transformed to a 0-100 scale with the higher values showing greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Jutras-Aswad, MD, Principal Investigator — CHUM
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No